CLINICAL TRIAL: NCT03104517
Title: CELLEBRATE: A Double-Blind, Randomized, Controlled Trial Comparing the Safety and Efficacy of AMDC-USR With Placebo in Female Subjects With Persistent or Recurrent Stress Urinary Incontinence Following Surgical Treatment
Brief Title: Autologous Muscle Derived Cells Compared to Placebo for Urinary Sphincter Repair in Post-surgical Female Stress Incontinence
Acronym: CELLEBRATE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-06
Expanded Access: NCT04661293 (Available)
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence; Urinary Stress Incontinence; Lower Urinary Tract Symptoms; Urinary Bladder; Urinary Tract Diseases; Bladder; Urinary Leak; Urine Leak; Bladder Leak; Urethra; Urethral Sphincter; Persistent Incontinence; Recurrent Incontinence; Incontinence Surgery; Sling Surgery; Stress Urinary Incontinence Surgery
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Lower Urinary Tract Symptoms; Urologic Diseases; Nocturnal Enuresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMDC-USR (iltamiocel) (Experimental): Autologous muscle-derived cells for urinary sphincter repair (AMDC-USR; generic name: iltamiocel) is the study product.
  Interventions: Biological: AMDC-USR (iltamiocel)
- Placebo (Placebo Comparator): Placebo control is the vehicle solution used for the study product.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AMDC-USR (iltamiocel) — Autologous Muscle Derived Cells for Urinary Sphincter Repair (generic name: iltamiocel)
  Arms: AMDC-USR (iltamiocel)
Other: Placebo — Placebo control is the vehicle solution used for the study product.
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of Autologous Muscle Derived Cells for Urinary Sphincter Repair (AMDC-USR; generic name: iltamiocel) compared to a placebo in the reduction of stress incontinence episode frequency in adult female patients with post-surgical persistent or recurrent stress urinary incontinence (SUI). Half of the participants will receive AMDC-USR (injections with cells) and the other half will receive placebo.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is the accidental loss of urine due to physical activity, such as laughing, coughing, or sneezing. Autologous Muscle Derived Cells for Urinary Sphincter Repair (AMDC-USR; generic name: iltamiocel) involves a medical procedure in which a participant's own muscle cells are collected, processed, and then injected into the tissues of the urinary passage.

This is a double-blind randomized study, which means neither the participant, nor the study doctor will know which treatment group the participant will be in. Participants who are randomly chosen to receive injection with placebo will have the option to receive an injection with their cells after completion of the blinded portion of their study participation (12 months).

ELIGIBILITY:
Inclusion Criteria:

* Adult female patient ≥ 18 years of age who has primary and moderate-to-severe symptoms of SUI for at least 6 months, as confirmed by patient medical history and clinical symptoms, including a focused incontinence evaluation.
* History of previous surgery for treatment of SUI. Previous surgery could include midurethral sling, retropubic suspension, or bladder neck sling. Bulking agents alone are not considered previous surgery for treatment of SUI.
* Must be willing and able to comply with the study procedures, be mentally competent and able to understand all study requirements, and must agree to read and sign the informed consent form prior to any study-related procedures.
* Must have completed 100% of the screening 3-day diary evening reports.

Exclusion Criteria:

* Patient has symptoms of only urge incontinence as confirmed by basic evaluation of etiology from a patient medical history, including a focused incontinence history.
* Patient has symptoms of mixed urinary incontinence where urge incontinence is the predominant factor.
* Patient has had stress urinary incontinence symptoms less than 6 months prior to signing the informed consent.
* Patient has not previously attempted conservative treatment prior to signing the informed consent. (Examples of conservative treatment include behavior modifications, bladder exercises, biofeedback, pelvic floor muscle therapy, etc.)
* Patient BMI ≥ 35.
* Patient routinely has more than 2 episodes of awakening to void during normal sleeping hours.
* If taking a medication known to affect lower urinary tract function, including but not limited to, anticholinergics, beta 3 adrenergic receptor agonists, tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitor (SNRI) or selective serotonin reuptake inhibitor (SSRI) antidepressants, diuretics, or alpha-adrenergic blockers, patient cannot be maintained on a stable dose and/or frequency of medication (including diuretics), cannot be maintained on a stable dose and/or frequency for at least 2 weeks prior to screening or is likely to change during the course of the study.
* History of cancer in pelvic organs, ureters, or kidneys.
* Patient is pregnant, lactating, or plans to become pregnant during the course of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of leaks due to stress incontinence episodes, as recorded in a diary | 12 months
  Stress leak frequency

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Kaufman, M.D., Ph.D., Principal Investigator — Vanderbilt University Medical Center, Department of Urologic Surgery
Locations (21):
- United States (20):
  - Arizona Urology Specialists, Tucson, Arizona
  - San Diego Clinical Trials, La Mesa, California
  - UCLA Women's Health Clinical Research Unit/Department of OBGYN, Los Angeles, California
  - Stanford Hospital and Clinics, Stanford, California
  - American Association of Female Pelvic Medicines Research Institute, Westlake Village, California
  - MedStar Georgetown Hospital Department of Urology, Washington D.C., District of Columbia
  - University of Kansas Health System, Kansas City, Kansas
  - Bennett Institute of Urogynecology and Incontinence, Grand Rapids, Michigan
  - University of New Mexico Women's Care Clinic, Albuquerque, New Mexico
  - AccuMed Research Associates, Garden City, New York
  - Northwell Health/The Arthur Smith Institute for Urology, Lake Success, New York
  - Columbia University Irving Medical Center, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Cleveland Clinic/Glickman Institute-Q10, Cleveland, Ohio
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Sanford Female Pelvic Medicine and Reconstructive Surgery Clinic, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Dept. of Urologic Surgery, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Cedar Health Research, Irving, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Derriford Hospital, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: https://www.suiclinicalstudy.com/ — https://www.suiclinicalstudy.com/